CLINICAL TRIAL: NCT02913781
Title: Polar Body Removal Before ICSI as a Method of Oocyte Activation in Previous Fertilization Failure Cases
Brief Title: Polar Body Removal Before ICSI for Oocyte Activation in Previous Fertilization Failure Cases
Acronym: PBRBICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Saad, Lecturer of Ob.&Gyn., Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hawaa-2
Record Dates: First submitted 2016-09-03; First posted 2016-09-26 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Fertilization
Keywords: Polar body removal; ICSI; Fertilization failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- polar body removal (Experimental): polar body removal by zona drilling with laser then suction by injecting pipette then ICSI procedure is done
  Interventions: Procedure: polar body removal using zona drilling by laser then suction by injecting pipette; Procedure: Classic ICSI

INTERVENTIONS:
Procedure: polar body removal using zona drilling by laser then suction by injecting pipette — zona drilling with laser followed by polar body removal then ICSI procedure
Procedure: Classic ICSI — Classic ICSI case was done be injecting sperm inside Oocyte while polar body is already existed at 6 or 12 O'clock position.

SUMMARY:
Cases which undergone ICSI before with failure of fertilization will do another ICSI cycle with removal of the polar body just before the ICSI procedure and sperm injection at the site of polar body removal. This study group will be evaluated with another group with the classic ICSI procedure

DETAILED DESCRIPTION:
Patients with previous fertilization failure will be divided into 2 groups:

Group 1 (control): Will undergo classic ICSI procedure in half the MII oocyte of the same case.

Group 2 (study group): The other half of the MII oocyte of the same case will undergo:

1. Polar body removal.
2. ICSI procedure with injection of the spermatozoon in the same zona opening (done by laser for polar body removal).

Results: Will be collected with evaluation of number of 2PN zygotes, Day 1, Day 2, Day 3, Day 5 embryos in all the cases.

ELIGIBILITY:
Inclusion Criteria:

* previous fertilization failure
* previous fertilization arrest

Exclusion Criteria:

* NO MII oocyte
* Refusal of the procedure by the couple

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
fertilization rate of the zygotes | 16-20 hours post ICSI
  fertilization check is done under inverted microscopy by 2PN check

SECONDARY OUTCOMES:
division rate of the embryos by the number of the blastomeres. | Day 2 & 3 & 5
  Detection of the number of the blastomeres and quality of the embryos under inverted microscopy. At day 5, detection of the rate of the blastocyst formation and quality of the embryos.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saad, Study Chair — Benha University
Locations (1):
- Banha University- Hawaa Fertility center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided